CLINICAL TRIAL: NCT03332654
Title: Prevalence and Risk Factors of Stress Urinary Incontinence in Women With Multiple Sclerosis
Brief Title: Stress Urinary Incontinence in Women With Multiple Sclerosis
Acronym: UROSEP
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-019
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Urinary Incontinence, Stress; Multiple Sclerosis
Keywords: Urinary Incontinence, Stress; Multiple Sclerosis; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Incontinence, Stress; Multiple Sclerosis; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis: Prevalence and risk factor of stress urinary incontinence in women with multiple sclerosis and included in the database over 15 years from December 1999 to June 2014, who had undergone a urodynamic test
  Interventions: Other: Determine prevalence of stress urinary incontinence

INTERVENTIONS:
Other: Determine prevalence of stress urinary incontinence

SUMMARY:
Objective: To report the prevalence and risk factors of stress urinary incontinence (SUI) and the prevalence of intrinsic sphincter deficiency in women with multiple sclerosis (MS). Methods: A retrospective study was conducted among Female patients with MS, followed for lower urinary tract symptoms (LUTS) during a 15-year period. Demographic data, MS history, expanded disability status scale (EDSS) score at the urodynamic visit, obstetrical past, birth weight, LUTS, and urodynamic findings were collected. SUI was defined as incontinence during cough, or any effort. A maximum urethral closure pressure less than 30 cm H2O defined intrinsic sphincter deficiency. Results: In total 363 women with a mean age of 46.7±10.8 years and a mean disease duration of 12.9±8.7 years were included. The incidence of relapsing remitting MS, a secondary progressive form, and a primary progressive form was 60.6%, 32.8%, and 6.6%, respectively. The prevalence of SUI was 31.4%. The prevalence of intrinsic sphincter deficiency was 1.4% and 0.8% of these patients had a SUI (P=0.300). In a multivariate analysis, women with a SUI had significantly higher birth weight (P=0.030), a pelvic organ prolapse (P=0.021), urgent urinary incontinence (P=0.006), a lower EDSS score (P=0.019), and a weaker containing effort (P<0.001). Conclusions: The prevalence of SUI in women with MS was 31.4%. This symptom could affect the quality of life of women with MS.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >18 years
* Multiple sclerosis
* Urodynamic test for lower urinary tract symptoms
* Followed in Saint Philibert Hospital between December 1999 to June 2014

Exclusion Criteria:

* Non confirmation of diagnosis of Multiple sclerosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All women aged >18 years with multiple sclerosis, who had undergone a urodynamic test for lower urinary tract symptoms were included
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Stress urinary incontinence | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Donzé, MD, Principal Investigator — GHICL